CLINICAL TRIAL: NCT02059759
Title: Immuno-modulation in Amyotrophic Lateral Sclerosis- a Phase II Study of Safety and Activity of Low Dose Interleukin-2
Acronym: IMODALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOCAL/2014/WC-01; 2014-001327-71 (EudraCT Number)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: low-dose interleukin 2
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — aldesleukin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Patients in this arm will receive sub-cutaneous injections of placebo (same vehicle as for experimental arms, and same volume) for 5 consecutive days at the beginning of three consecutive months (a total of 15 injections, 5 per month for 3 months).
  Intervention: Placebo
  Interventions: Drug: Placebo
- 1.0 IL-2 (Experimental): Patients in this arm will receive sub-cutaneous injections corresponding to 1.0 MIU of IL-2 per injection for 5 consecutive days at the beginning of three consecutive months (a total of 15 injections, 5 per month for 3 months).
  Intervention: 1.0 MIU IL-2 per day
  Interventions: Drug: 1.0 MIU IL-2 per day
- 2.0 IL-2 (Experimental): Patients in this arm will receive sub-cutaneous injections corresponding to 2.0 MIU of IL-2 per injection for 5 consecutive days at the beginning of three consecutive months (a total of 15 injections, 5 per month for 3 months).
  Intervention: 2.0 MIU IL-2 per day
  Interventions: Drug: 2.0 MIU IL-2 per day

INTERVENTIONS:
Drug: Placebo — Patients in this arm will receive sub-cutaneous injections of placebo (same vehicle as for experimental arms, and same volume) for 5 consecutive days at the beginning of three consecutive months (a total of 15 injections, 5 per month for 3 months).
  Arms: Placebo
Drug: 1.0 MIU IL-2 per day — Patients in this arm will receive sub-cutaneous injections corresponding to 1.0 MIU of IL-2 per injection for 5 consecutive days at the beginning of three consecutive months (a total of 15 injections, 5 per month for 3 months).
  Other Names: Aldesleukine; Proleukin
  Arms: 1.0 IL-2
Drug: 2.0 MIU IL-2 per day — Patients in this arm will receive sub-cutaneous injections corresponding to 2.0 MIU of IL-2 per injection for 5 consecutive days at the beginning of three consecutive months (a total of 15 injections, 5 per month for 3 months).
  Other Names: Aldesleukine; Proleukin
  Arms: 2.0 IL-2

SUMMARY:
The primary objective is to evaluate in ALS patients the regulatory T cell early response to two low-doses of IL-2 at 1 and 2 MIU per day after one course of 5 consecutive days comparatively to placebo.

DETAILED DESCRIPTION:
This is a phase II study on ld-IL-2 as a therapeutic agent for ALS which aims at defining the activity and safety of a range a doses for subsequent use of the best dose in a phase II/III trial. For ethical reasons, ld-IL-2 must be tested as an add-on therapy to riluzole hence all patients will need to be treated with riluzole for at least three months prior to entry. A randomized (1:1:1), placebo-controlled, double-blind, parallel group trial will be carried out to assess ld-IL-2 activity on regulatory T cells and immuno-inflammatory markers in ALS patients treated for 3 months (5 days every four weeks repeated three times).

The secondary objectives of this study are:

A. To evaluate maintenance of Tcell response after three repeated 5-day courses at one course every four weeks for 12 weeks.

B. To evaluate the safety of ld-IL-2 therapy in an ALS population, with an overall follow-up of 6 months (up to 15 weeks after last administration); C. To evaluate functional changes throughout the study; D. To evaluate changes in other pre-defined blood cytology parameters, and a blood biomarker for axonal damage.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been correctly informed
* The patient must have given his/her informed and signed consent.
* The patient must be insured or beneficiary of a health insurance plan.
* The patient is at least 18 years old and less than 75 years old
* Probable, or laboratory-supported probable or definite ALS as defined by El Escorial Revised ALS diagnostic criteria (according to Airlie House Conference 1988)
* Stable on riluzole treatment for more than 3 months with liver function test results < 2ULN
* Disease duration ≤ 5 years
* Vital capacity ≥ 70% of normal
* Ability to swallow without the requirement for nasogastric or PEG feeding
* Agreement for patient to use an adequate method of contraception throughout the study and for 2 weeks after post study visit
* The patient is available and willing to participate in seven study visits occurring at the CHU within the next six months

Exclusion Criteria:

* The patient is participating in another interventional study
* Within the past three months, the patient has participated in another interventional
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The patient is an adult under guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Other life threatening disease
* Presence of contra-indicated concomitant treatments or with potential neuroprotective benefit (see section 11.2 of the protocol)
* Presence of tracheostomy or non-invasive ventilation
* Use of Percutaneous endoscopic gastrostomy (PEG) or nasogastric tube
* Presence of clinical infection (treated or untreated)
* Positive serology for CMV, EBV (confirmed by viral load), or HIV
* Vaccination within 8 weeks prior to first experimental dosing
* Other disease precluding functional assessments
* Cancer within the past 5 years (except stable non-metastatic basal cell skin carcinoma or in situ carcinoma of the cervix)
* Severe cardiac or pulmonary disease
* Documented auto-immune disorders except asymptomatic Hashimoto thyroiditis
* Women of child bearing age without contraception or pregnant or breast feeding
* Any clinically significant laboratory abnormality (excepting cholesterol, triglyceride and glucose)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
CD4+ CD25+ CD127- FoxP3+(Treg) cells: change in percentage of total lymphocytes | Day 8
  Treg refers to regulatory T cells

SECONDARY OUTCOMES:
Presence/absence of specific, pre-defined adverse events. | Day 1
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 2
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 3
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 4
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 5
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 6
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 7
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 8
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 29
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 30
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 31
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 32
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 33
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 34
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 35
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 36
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 57
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 58
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 59
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 60
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 61
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 62
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 63
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of specific, pre-defined adverse events. | Day 64
  The pre-defined events include: injection site reaction, flu like syndrome, fatigue, gastro-intestinal signs, allergic signs.
Presence/absence of abnormal vital signs | Day 1
  (based on a systematic check of vital signs: pulse, blood pressure, oxymetry, temperature)
Presence/absence of abnormal vital signs | Day 8
  (based on a systematic check of vital signs: pulse, blood pressure, oxymetry, temperature)
Presence/absence of abnormal vital signs | Day 29
  (based on a systematic check of vital signs: pulse, blood pressure, oxymetry, temperature)
Presence/absence of abnormal vital signs | Day 57
  (based on a systematic check of vital signs: pulse, blood pressure, oxymetry, temperature)
Presence/absence of abnormal vital signs | Day 64
  (based on a systematic check of vital signs: pulse, blood pressure, oxymetry, temperature)
Presence/absence of abnormal vital signs | Week 13
  (based on a systematic check of vital signs: pulse, blood pressure, oxymetry, temperature)
Presence/absence of abnormal vital signs | Week 25
  (based on a systematic check of vital signs: pulse, blood pressure, oxymetry, temperature)
MedDRA classification of all adverse events throughout the study | Week 25
  MedDRA refers to "Medical Dictionary for Regulatory Activities"
Thyroid function: blood T4 | Baseline (day 0 to day -15)
Thyroid function: blood T4 | Week 13
Thyroid function: blood TSH | Baseline (day 0 to day -15)
Thyroid function: blood TSH | Week 13
Presence/absence of clinically significant abnormality on a lung x-ray | Baseline (day 0 to day -15)
Presence/absence of clinically significant abnormality on a lung x-ray | Week 13
Presence/absence of clinically significant abnormality on an electrocardiogram | Baseline (day 0 to day -15)
Presence/absence of clinically significant abnormality on an electrocardiogram | Week 13
Presence/absence of a clinically significant abnormality among routine laboratory tests | Day 1
  The routine blood tests considered are:
  * haemogram (hemoglobin, hematocrit, red blood cell count, white blood cell count, leukocyte formula, platelets, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration )
  * blood biochemistry (ionogram, urea, creatinine, glucose, C reactive protein, procalcitonin, protein, albumin)
  * liver function panel (aspartate transaminase, alanine transaminase, gamma-glutamyl transpeptidase, bilirubin)
  * iron metabolism (iron, ferritin, transferrin)
Presence/absence of a clinically significant abnormality among routine laboratory tests | Day 8
  The routine blood tests considered are:
  * haemogram (hemoglobin, hematocrit, red blood cell count, white blood cell count, leukocyte formula, platelets, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration)
  * blood biochemistry (ionogram, urea, creatinine, glucose, C reactive protein, procalcitonin, protein, albumin)
  * liver function panel (aspartate transaminase, alanine transaminase, gamma-glutamyl transpeptidase, bilirubin)
  * iron metabolism (iron, ferritin, transferrin)
Presence/absence of a clinically significant abnormality among routine laboratory tests | Day 29
  The routine blood tests considered are:
  * haemogram (hemoglobin, hematocrit, red blood cell count, white blood cell count, leukocyte formula, platelets, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration)
  * blood biochemistry (ionogram, urea, creatinine, glucose, C reactive protein, procalcitonin, protein, albumin)
  * liver function panel (aspartate transaminase, alanine transaminase, gamma-glutamyl transpeptidase, bilirubin)
  * iron metabolism (iron, ferritin, transferrin)
Presence/absence of a clinically significant abnormality among routine laboratory tests | Day 57
  The routine blood tests considered are:
  * haemogram (hemoglobin, hematocrit, red blood cell count, white blood cell count, leukocyte formula, platelets, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration)
  * blood biochemistry (ionogram, urea, creatinine, glucose, C reactive protein, procalcitonin, protein, albumin)
  * liver function panel (aspartate transaminase, alanine transaminase, gamma-glutamyl transpeptidase, bilirubin)
  * iron metabolism (iron, ferritin, transferrin)
Presence/absence of a clinically significant abnormality among routine laboratory tests | Day 64
  The routine blood tests considered are:
  * haemogram (hemoglobin, hematocrit, red blood cell count, white blood cell count, leukocyte formula, platelets, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration)
  * blood biochemistry (ionogram, urea, creatinine, glucose, C reactive protein, procalcitonin, protein, albumin)
  * liver function panel (aspartate transaminase, alanine transaminase, gamma-glutamyl transpeptidase, bilirubin)
  * iron metabolism (iron, ferritin, transferrin)
Presence/absence of a clinically significant abnormality among routine laboratory tests | Week 13
  The routine blood tests considered are:
  * haemogram (hemoglobin, hematocrit, red blood cell count, white blood cell count, leukocyte formula, platelets, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration)
  * blood biochemistry (ionogram, urea, creatinine, glucose, C reactive protein, procalcitonin, protein, albumin)
  * liver function panel (aspartate transaminase, alanine transaminase, gamma-glutamyl transpeptidase, bilirubin)
  * iron metabolism (iron, ferritin, transferrin)
Presence/absence of a clinically significant abnormality among routine laboratory tests | Week 25
  The routine blood tests considered are:
  * haemogram (hemoglobin, hematocrit, red blood cell count, white blood cell count, leukocyte formula, platelets, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration)
  * blood biochemistry (ionogram, urea, creatinine, glucose, C reactive protein, procalcitonin, protein, albumin)
  * liver function panel (aspartate transaminase, alanine transaminase, gamma-glutamyl transpeptidase, bilirubin)
  * iron metabolism (iron, ferritin, transferrin)
Vital capacity (% of normal) | Baseline (day 0 to day -15)
  This is a measure of respiratory function.
Vital capacity (% of normal) | Day 1
  This is a measure of respiratory function.
Vital capacity (% of normal) | Week 13
  This is a measure of respiratory function.
Vital capacity (% of normal) | Week 25
  This is a measure of respiratory function.
The ALSFRS Questionnaire | Day 1
The ALSFRS Questionnaire | Day 29
The ALSFRS Questionnaire | Day 57
The ALSFRS Questionnaire | Week 13
The ALSFRS Questionnaire | Week 25
Tregs (absolute number and % CF4+ cells) | Day 1
Tregs (absolute number and % CF4+ cells) | Day 8
Tregs (absolute number and % CF4+ cells) | Day 57
Tregs (absolute number and % CF4+ cells) | Day 64
Tregs (absolute number and % CF4+ cells) | Week 13
Tregs (absolute number and % CF4+ cells) | Week 25
Total lymphocyte number | Day 1
Total lymphocyte number | Day 8
Total lymphocyte number | Day 57
Total lymphocyte number | Day 64
Total lymphocyte number | Week 13
Total lymphocyte number | Week 25
CD56+(NK), CD19+(B), CD3+, CD4+, CD8+ cell populations: numbers and percentages of total lymphocytes | Day 1
CD56+(NK), CD19+(B), CD3+, CD4+, CD8+ cell populations: numbers and percentages of total lymphocytes | Day 8
CD56+(NK), CD19+(B), CD3+, CD4+, CD8+ cell populations: numbers and percentages of total lymphocytes | Day 57
CD56+(NK), CD19+(B), CD3+, CD4+, CD8+ cell populations: numbers and percentages of total lymphocytes | Day 64
CD56+(NK), CD19+(B), CD3+, CD4+, CD8+ cell populations: numbers and percentages of total lymphocytes | Week 13
CD56+(NK), CD19+(B), CD3+, CD4+, CD8+ cell populations: numbers and percentages of total lymphocytes | week 25
effector T cells: number and % of CD4 cells | Day 1
  This is measured as CD4+ lymphocytes minus regulatory T cells
effector T cells: number and % of CD4 cells | Day 8
  This is measured as CD4+ lymphocytes minus regulatory T cells
effector T cells: number and % of CD4 cells | Day 57
  This is measured as CD4+ lymphocytes minus regulatory T cells
effector T cells: number and % of CD4 cells | Day 64
  This is measured as CD4+ lymphocytes minus regulatory T cells
effector T cells: number and % of CD4 cells | Week 13
  This is measured as CD4+ lymphocytes minus regulatory T cells
effector T cells: number and % of CD4 cells | Week 25
  This is measured as CD4+ lymphocytes minus regulatory T cells
Phosphorylated neurofilament heavy protein (pNfH) levels in serum | day 1
Light chain neurofilament levels in serum | Day 1
Light chain neurofilament levels in serum | Week 13

OTHER OUTCOMES:
Age (years) | Baseline
Sex (male/female) | Baseline
Body mass index (kg/m^2) | Baseline
Disease duration from date of first symptoms (fatigue, weakness) | Baseline
The patient's current Riluzole posology | Baseline to week 25
The patient's currentposology for other concomitant treatments | Baseline to week 25
Description of concomitant treatments, if any | Throughout study, up to 25 weeks
Routine serology results dating to within the last 30 days: HIV-1 (positive/negative ?) | Baseline
Routine serology results dating to within the last 30 days: Epstein Barr Virus (positive/negative ?) | Baseline
Routine serology results dating to within the last 30 days: cytomegalovirus (positive/negative ?) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raul Juntas-Morales, MD, Study Director — CHRU de Montpellier
Locations (1):
- CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier, France

REFERENCES:
- [Result] Camu W, Mickunas M, Veyrune JL, Payan C, Garlanda C, Locati M, Juntas-Morales R, Pageot N, Malaspina A, Andreasson U, Kirby J, Suehs C, Saker S, Masseguin C, De Vos J, Zetterberg H, Shaw PJ, Al-Chalabi A, Leigh PN, Tree T, Bensimon G. Repeated 5-day cycles of low dose aldesleukin in amyotrophic lateral sclerosis (IMODALS): A phase 2a randomised, double-blind, placebo-controlled trial. EBioMedicine. 2020 Sep;59:102844. doi: 10.1016/j.ebiom.2020.102844. Epub 2020 Jul 7. PMID 32651161